CLINICAL TRIAL: NCT04681495
Title: Translating an In-Person Brief, Bystander Bullying Intervention (STAC) to a Technology-Based Intervention
Acronym: STAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Boise State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 325; 1R41MD014943-01 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Bullying of Child; Bullying
Keywords: Bullying; Bullying Prevention; Technology
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usability of Bullying Prevention Online Application (Other): This intervention has a single arm. It consists of conducting focus groups and usability testing of a bullying prevention online application for middle-school-aged students.
  Interventions: Behavioral: STAC

INTERVENTIONS:
Behavioral: STAC — STAC is a brief, stand-alone bullying bystander intervention for middle school students, to reduce bullying and mental health risks for bystanders. The primary outcome will be showing usability for the technology-based program (STAC-T) prototype.

SUMMARY:
School interventions to reduce bullying can be effective but also require substantial time and resources. Online technologies have the potential to deliver effective bullying interventions to a large number of middle schools for less cost. The feasibility of delivering the effective STAC bullying intervention through a mobile web app will be tested using a needs analysis with school administrators, focus groups with middle school students, and development and usability testing of a prototype.

DETAILED DESCRIPTION:
While studies support the efficacy of comprehensive, school-wide interventions in reducing bullying, these types of programs can require significant time and financial resources for implementation, resulting in barriers to providing school-based bullying prevention, especially in low-income and rural communities. Additionally, although training bystanders to act as "defenders" on behalf of targets of bullying is an important intervention component, few programs include this as part of their comprehensive strategy. Brief programs that focus on bystander training and require fewer resources are needed to reduce bullying and its negative consequences. The PI (Dr. Midgett) developed STAC, a brief, stand-alone bullying bystander intervention for middle school students, to reduce bullying and mental health risks for bystanders. Brief, in-person programs, however, still pose implementation barriers such as training school personnel, providing external support, and not allowing for large groups of students to be trained at the same time. For this project, we propose to develop a technology-based STAC intervention (STAC-T) that will allow students to customize their experience by selecting avatars and bullying scenarios based on our previous studies conducted in a range of middle schools, including those in low-income and rural communities. The innovative, user-centered design proposed will be inherently sensitive to cultural needs of students and identify personally-appropriate strategies. The specific aims of this application include conducting a needs analysis to determine product need, building a system prototype leveraging prior work and expertise of an external advisory board, and usability and effectiveness testing with middle school students and stakeholders to evaluate feasibility. This proposal is designed to document proof of concept and finalizing design and content of the system which will be developed and tested in a subsequent randomized controlled trial. The technology-based platform will increase the overall reach, impact, and sustainability of the STAC intervention for bullying prevention. It will substantially reduce cost to increase reach and its interactivity and algorithms can tailor program content to adapt it further for students attending low-income and rural schools. Thus, this low-cost, easy to disseminate technology-based bullying bystander intervention has the potential to have a substantial impact on the problem of bullying and the negative associated consequences for both students who are targets and bystanders in middle school when the problem of bullying peaks. There is a large market for the STAC-T intervention with approximately 100,000 public and private schools with middle-school grades in the United States. Globally, the online education market is growing at 10% a year and the digital health market exceeds $220 billion annually.

ELIGIBILITY:
Inclusion Criteria (Students):

* Enrolled in grades 6, 7, 8, or 9 in a middle/junior high school in Idaho.
* Have a desire to make a positive difference at school, be mature, and have ability to positively engage socially with peers and adults as judged by school personnel.
* Speaks and reads English
* Parent consents and students assents for participation

Inclusion Criteria (School Personnel)

* Employed in a middle/junior high school in Idaho with grades 6, 7, 8, and/or 9.
* Employed as a principal, teacher, or school counselor
* Speaks and reads English
* Consents to participate

Exclusion Criteria (Students):

* Participated in a previous study on STAC
* Speaks and reads only a language other than English
* Does not consent/assent

Exclusion Criteria (School Personnel):

* Participated in a previous study on STAC
* Speaks and reads only a language other than English
* Does not consent/assent

Ages: 11 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
System Usability Questionnaire | The SUS will be completed one time immediately following usability testing. The usability testing will last one hour and will be conducted in months 9 through 11 of the study..
  Participant perspective of program feasibility and bullying prevention promotion. The System Usability Scale (SUS) is a reliable tool for measuring the usability of technologies. It consists of a 10-item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average.

CONTACTS AND LOCATIONS:
Overall Officials: Aida Midgett, PhD, LPC, Principal Investigator — Boise State University
Locations (2):
- United States (2):
  - Klein Buendel, Inc, Golden, Colorado
  - Boise State University, Boise, Idaho

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Midgett A, Doumas DM, Myers VH, Moody S, Doud A. Technology-Based Bullying Intervention for Rural Schools: Perspectives on Needs, Challenges, and Design. Rural Ment Health. 2021 Jan;45(1):14-30. doi: 10.1037/rmh0000151. PMID 33777286
- [Derived] Doumas DM, Midgett A, Myers V, Buller MK. Usability of a Technology-Based Bystander Bullying Intervention for Middle School Students in Rural, Low-Income Communities: Mixed Methods Study. JMIR Form Res. 2021 Oct 26;5(10):e32382. doi: 10.2196/32382. PMID 34582355